CLINICAL TRIAL: NCT02394119
Title: Ofatumumab Versus Rituximab in Children With Steroid and Calcineurin Inhibitor-dependent Idiopathic Nephrotic Syndrome: an Open-label, Randomized, Controlled, Superiority Trial.
Brief Title: Ofatumumab Versus Rituximab in Children With Steroid and Calcineurin Inhibitor Dependent Idiopathic Nephrotic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Giannina Gaslini (Other)
Responsible Party: Principal Investigator, Gian Marco Ghiggeri MD, PhD, MD, director of Nephrology, Dialysis and Transplantation Unit, Istituto Giannina Gaslini
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OFA2
Record Dates: First submitted 2015-03-06; First posted 2015-03-20 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Nephrotic Syndrome
MeSH Terms: conditions — Nephrotic Syndrome | interventions — ofatumumab; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ofatumumab (Experimental): * Drug Name: Ofatumumab
  * Why: Anti-body/antigen interaction results in cell apoptosis and reduced CD20 positive cell related activities
  * Procedures: methylprednisolone 2 mg/kg infused in 30' IV diluted in 100 ml of normal saline (NaCl 0,9%); oral paracetamol 15 mg/kg ; cetirizine 0,4 mg/kg IV infused slowly in 5 ml of normal saline (NaCl 0,9%) prior to Ofatumumab infusion to reduce common reactions
  * How: Ofatumumab IV: 1500 mg/1.73m2 at 12 ml/hour in the first 30'. Thereafter, the infusion rate can be doubled every 30 minutes up to a maximum of 200 ml/hour.
  * When and how much: once; diluted in 1000 ml of normal saline.
  Interventions: Drug: Ofatumumab
- Rituximab (Active Comparator): * Drug Name: Rituximab (RTX)
  * Why: Anti-body/antigen interaction results in cell apoptosis and reduced CD20 positive cell related activities
  * Procedures: the same as for Ofatumumab Arm
  * How: Rituximab IV: 375 mg/m2; for dosage between 100 and 250 mg RTX will be diluted in 100 ml of normal saline and administered at 2 ml/h for the first 30'; 3 ml/h for the second 30'; 6 ml/h for the third 30'; 15 ml/h until the end. For dosage between 260 and 500 mg RTX will be diluted in 250 ml of normal saline and administered at 6 ml/h for the first 30'; 9 ml/h for the second 30'; 18 ml/h for the third 30'; 36 ml/h until the end. For dosage between 510 and 1000 mg RTX will be diluted in 500 ml of normal saline and administered at 9 ml/h for the first 30'; thereafter, the infusion rate can be doubled every 30 minutes up to a maximum of 72 ml/h.
  * When and how much: once; diluted in 100/250/500 ml of normal saline for dosage respectively between 100-250 mg, 260-500 mg, 510-1000 mg.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Ofatumumab — 1500 mg/1.73m2, administered once diluted in 1000 ml of normal saline
  Other Names: Arzerra
  Arms: Ofatumumab
Drug: Rituximab — 375 mg/m2, administered once diluted in 100/250/500 ml of normal saline for dosage respectively between 100-250 mg, 260-500 mg, 510-1000 mg.
  Other Names: Mabthera
  Arms: Rituximab

SUMMARY:
Open-label, two-parallel-arm, controlled randomized clinical trial testing the superiority of Ofatumumab over Rituximab in maintaining steroid- and calcineurin-inhibitor-free disease remission in SD-INS.

Eligible participants will enter a 1-month run-in period, during which instruction on urine collection and dipstick readings will be carefully reviewed, compliance assessed, and therapy with RAS inhibitors withdrawn and, in hypertensive children replaced by other anti-hypertensive drug.

After run-in period, children will be randomized to either the intervention arm (Ofatumumab) or the comparator arm (Rituximab).

After infusion of intervention or comparator, steroids will be maintained at initial dose for 30 days and then tapered off by 0.3 mg/kg per week until complete withdrawal.

One week after the steroid withdrawal calcineurin inhibitors will be decreased by 50% and withdrawn within 2 additional weeks.

All patients will be followed for up to 24 months. In case of relapses during the study (see outcome section for definition) patients will be treated with 60 mg/m2of prednisone p.o. in order to achieve remission. At remission, patients will be treated with another infusion of either Oftumumab or Rituximab, according to the initial randomization.

After infusion of intervention or comparator, steroids will be maintained at initial dose for 30 days and then tapered off by 0.3 mg/kg per week until complete withdrawal.

One week after the steroid withdrawal calcineurin-inhibitors will be decreased by 50% and withdrawn within 2 additional weeks. This strategy will be repeated to treat full relapses during the study.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion into this study, participants will have to fulfill the following criteria:

* To be in complete disease remission
* Drug dependence: remission has to be maintained with both steroids and CNI steroid dependence is defined by two consecutive relapses during corticosteroid therapy or within 14 days of ceasing therapy. CNI (cyclosporine/tacrolimus) dependence is defined by presence of relapse at discontinuation.
* Ability to provide consent and assent: parents'/guardian's written informed consent, and child's assent given before any study-related procedure not part of the subject's normal medical care, with the understanding that consent may be withdrawn by the subject at any time without prejudice to his or her future medical care.
* Age between 2 and 24 years

Exclusion Criteria:

Children will be excluded if any of the following criteria apply:

* Positivity to autoimmunity tests (ANA, nDNA, ANCA)
* Reduction of C3 levels.
* eGFR<90/ml/min/1,73 m2 valuated according to revised Bedside Schwartz Formula for patients between 2 and 17 years and with CKD-EPI Creatinine 2009 Equation for 18 years old patients.
* Pregnancy
* Neoplasm
* Infections: previous or actual HBV (with HBeAb positivity) or HCV infection
* CD20 B lymphocytes count <2,5%
* Treatment with Rituximab or cyclophosphamide in the last 6 months

Ages: 2 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Actual)
Dates: Start 2015-06; Primary Completion 2018-06 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Risk of relapse | 12 months
  The primary endpoints will be risk of relapse at 12 months without steroid or calcineurin-inhibitors. Relapse is defined by uPCR ≥2000 mg/g (≥ 200 mg/mmol) or > 3+ protein on urine dipstick for 3 consecutive days (KDIGO Clinical Practice Guideline for Glomerulonephritis, Kidney International Supplement, 2012 2, 163-171).

SECONDARY OUTCOMES:
Amount of steroids required to maintain complete disease remission | 6 and 24 months after Ofatumumab or Rituximab pulse
  Complete remission is defined by uPCR <200 mg/g (<20 mg/mmol) or o1+ of protein on urine dipstick for 3 consecutive days (KDIGO Clinical Practice Guideline for Glomerulonephritis, Kidney International Supplement, 2012 2, 163-171).
Adverse events | At 1, 3, 6, 9 ,12, 15, 18, 21 and 24 months after drug infusion, during protocol visits.
  Measurement of frequency and severity of adverse events due to drug infusion
Abnormal laboratory values | At 1, 3, 6, 9 ,12, 15, 18, 21 and 24 months after drug infusion, during protocol visits.
  Record of abnormal values in biochemical tests and hematology assessments due to drug infusion

CONTACTS AND LOCATIONS:
Overall Officials: Gianmarco Ghiggeri, MD, Principal Investigator — Istituto Giannina Gaslini
Locations (1):
- IRCCS Istituto Giannina Gaslini, Genoa, Italy/GE, Italy

REFERENCES:
- [Background] McEnery PT, Strife CF. Nephrotic syndrome in childhood. Management and treatment in patients with minimal change disease, mesangial proliferation, or focal glomerulosclerosis. Pediatr Clin North Am. 1982 Aug;29(4):875-94. No abstract available. PMID 7050865
- [Background] Hodson EM, Knight JF, Willis NS, Craig JC. Corticosteroid therapy for nephrotic syndrome in children. Cochrane Database Syst Rev. 2005 Jan 25;(1):CD001533. doi: 10.1002/14651858.CD001533.pub3. PMID 15674881
- [Background] Ravani P, Rossi R, Bonanni A, Quinn RR, Sica F, Bodria M, Pasini A, Montini G, Edefonti A, Belingheri M, De Giovanni D, Barbano G, Degl'Innocenti L, Scolari F, Murer L, Reiser J, Fornoni A, Ghiggeri GM. Rituximab in Children with Steroid-Dependent Nephrotic Syndrome: A Multicenter, Open-Label, Noninferiority, Randomized Controlled Trial. J Am Soc Nephrol. 2015 Sep;26(9):2259-66. doi: 10.1681/ASN.2014080799. Epub 2015 Jan 15. PMID 25592855
- [Background] Iijima K, Sako M, Nozu K, Mori R, Tuchida N, Kamei K, Miura K, Aya K, Nakanishi K, Ohtomo Y, Takahashi S, Tanaka R, Kaito H, Nakamura H, Ishikura K, Ito S, Ohashi Y; Rituximab for Childhood-onset Refractory Nephrotic Syndrome (RCRNS) Study Group. Rituximab for childhood-onset, complicated, frequently relapsing nephrotic syndrome or steroid-dependent nephrotic syndrome: a multicentre, double-blind, randomised, placebo-controlled trial. Lancet. 2014 Oct 4;384(9950):1273-81. doi: 10.1016/S0140-6736(14)60541-9. Epub 2014 Jun 22. PMID 24965823
- [Background] Ravani P, Magnasco A, Edefonti A, Murer L, Rossi R, Ghio L, Benetti E, Scozzola F, Pasini A, Dallera N, Sica F, Belingheri M, Scolari F, Ghiggeri GM. Short-term effects of rituximab in children with steroid- and calcineurin-dependent nephrotic syndrome: a randomized controlled trial. Clin J Am Soc Nephrol. 2011 Jun;6(6):1308-15. doi: 10.2215/CJN.09421010. Epub 2011 May 12. PMID 21566104
- [Background] Basu B. Ofatumumab for rituximab-resistant nephrotic syndrome. N Engl J Med. 2014 Mar 27;370(13):1268-70. doi: 10.1056/NEJMc1308488. No abstract available. PMID 24670185
- [Background] Robak T. Ofatumumab, a human monoclonal antibody for lymphoid malignancies and autoimmune disorders. Curr Opin Mol Ther. 2008 Jun;10(3):294-309. PMID 18535937
- [Background] Magnasco A, Ravani P, Edefonti A, Murer L, Ghio L, Belingheri M, Benetti E, Murtas C, Messina G, Massella L, Porcellini MG, Montagna M, Regazzi M, Scolari F, Ghiggeri GM. Rituximab in children with resistant idiopathic nephrotic syndrome. J Am Soc Nephrol. 2012 Jun;23(6):1117-24. doi: 10.1681/ASN.2011080775. Epub 2012 May 10. PMID 22581994
- [Background] Ravani P, Ponticelli A, Siciliano C, Fornoni A, Magnasco A, Sica F, Bodria M, Caridi G, Wei C, Belingheri M, Ghio L, Merscher-Gomez S, Edefonti A, Pasini A, Montini G, Murtas C, Wang X, Muruve D, Vaglio A, Martorana D, Pani A, Scolari F, Reiser J, Ghiggeri GM. Rituximab is a safe and effective long-term treatment for children with steroid and calcineurin inhibitor-dependent idiopathic nephrotic syndrome. Kidney Int. 2013 Nov;84(5):1025-33. doi: 10.1038/ki.2013.211. Epub 2013 Jun 5. PMID 23739238
- [Derived] Larkins NG, Hahn D, Liu ID, Willis NS, Craig JC, Hodson EM. Non-corticosteroid immunosuppressive medications for steroid-sensitive nephrotic syndrome in children. Cochrane Database Syst Rev. 2024 Nov 8;11(11):CD002290. doi: 10.1002/14651858.CD002290.pub6. PMID 39513526
- [Derived] Ravani P, Colucci M, Bruschi M, Vivarelli M, Cioni M, DiDonato A, Cravedi P, Lugani F, Antonini F, Prunotto M, Emma F, Angeletti A, Ghiggeri GM. Human or Chimeric Monoclonal Anti-CD20 Antibodies for Children with Nephrotic Syndrome: A Superiority Randomized Trial. J Am Soc Nephrol. 2021 Oct;32(10):2652-2663. doi: 10.1681/ASN.2021040561. Epub 2021 Sep 20. PMID 34544820
- [Derived] Ravani P, Bonanni A, Ghiggeri GM. Randomised controlled trial comparing ofatumumab to rituximab in children with steroid-dependent and calcineurin inhibitor-dependent idiopathic nephrotic syndrome: study protocol. BMJ Open. 2017 Mar 17;7(3):e013319. doi: 10.1136/bmjopen-2016-013319. PMID 28314744